CLINICAL TRIAL: NCT07105176
Title: A Phase Ib Single-arm Clinical Study of HS-IT101 Injection for Advanced NSCLC
Brief Title: HS-IT101 Injection for Advanced NSCLC
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qingdao Sino-Cell Biomedicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-IT101ST01-Ⅰ b-02
Record Dates: First submitted 2025-07-22; First posted 2025-08-05 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07

CONDITIONS: Advanced Non-Small Cell Lung Cancer
MeSH Terms: interventions — Cyclophosphamide; fludarabine; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HS-IT101 monotherapy (Experimental): TIL Injection administered by intravenous infusion over 30-60 minutes.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: IL-2 (interleukin 2); Drug: HS-IT101 monotherapy

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide administered via intravenous infusion once daily for 3 consecutive days.
Drug: Fludarabine — Fludarabine is administered once daily via intravenous infusion for 4 consecutive days.
Drug: IL-2 (interleukin 2) — IL-2 administered subcutaneously once daily. Dosing may be adjusted based on subject tolerance, including modifications to dose quantity, administration frequency, or complete treatment discontinuation, with a maximum treatment duration of 3 days.
Drug: HS-IT101 monotherapy — TIL Injection administered by intravenous infusion over 30-60 minutes.

SUMMARY:
An Open-Label, Single-Arm Phase Ib Clinical Trial Evaluating the Safety, Tolerability, and Preliminary Efficacy of HS-IT101 Injection in Subjects with Advanced NSCLC.

DETAILED DESCRIPTION:
A Single-Arm, Open-Label, Interventional Study Evaluating Adoptive Cell Therapy (ACT) with Autologous Tumor-Infiltrating Lymphocytes (HS-IT101) Following Lymphodepleting Conditioning with Fludarabine and Cyclophosphamide, Followed by IL-2 in Patients with Advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70 years (inclusive).

Diagnosis:

Histologically/cytologically confirmed advanced, recurrent, or metastatic non-small cell lung cancer (NSCLC) .

Tumor Sampling:

≥1 lesion untreated with radiotherapy/local therapy within 28 days for TIL preparation (tissue weight ≥0.050 g).

Target Lesion:

≥1 measurable lesion per RECIST v1.1, untreated with radiotherapy/local therapy (unless treatment occurred >28 days before sampling with documented progression).

Performance Status: ECOG score ≤1. Survival: Life expectancy ≥3 months.

Organ Function:

Hematology: ANC ≥1.5×10⁹/L, PLT ≥90×10⁹/L, HGB ≥90 g/L (no transfusion/erythropoietin within 14 days).

Liver: ALT/AST ≤2.5×ULN (≤5×ULN if liver metastases); TBil ≤1.5×ULN (≤3×ULN for Gilbert syndrome).

Kidney: Serum Cr ≤1.5×ULN or Ccr ≥60 mL/min (Cockcroft-Gault formula). Coagulation: APTT ≤1.5×ULN; INR/PT ≤1.5×ULN.

Cardiac Function:

LVEF ≥50% by echocardiography; QTcF ≤470 ms (Fridericia formula: QTcF = QT/RR⁰·³³).

Baseline SpO₂ >91% (room air). Note: If QTcF is abnormal initially, repeat twice at ≥5-minute intervals and use mean value for eligibility.

Toxicity Recovery: All treatment-related adverse events resolved to CTCAE v5.0 ≤Grade 1 (except alopecia/non-risk toxicities per investigator) before tumor sampling.

Contraception: Effective non-pharmacological contraception from informed consent until 1 year post-TIL infusion.

Compliance: Capable of understanding the trial, voluntarily signing informed consent, and adhering to protocol visits/procedures.

Exclusion Criteria:

* Severe Hypersensitivity: History of severe hypersensitivity to drugs used in the study (including but not limited to cyclophosphamide, fludarabine, IL-2, gentamicin, amphotericin B, or components of TIL infusion).

Uncontrolled Comorbidities:

Poorly controlled hypertension (resting SBP ≥160 mmHg or DBP ≥100 mmHg despite medication).

Congestive heart failure (NYHA Class III/IV).

Cardiovascular Events (within 6 months):

Deep vein thrombosis, pulmonary embolism, myocardial infarction, severe/unstable arrhythmia, angina, PCI, ACS, CABG, stroke, TIA, or cerebral embolism.

Active Autoimmune Disease:

Requires systemic therapy during the study period (Exceptions: Eczema, vitiligo, psoriasis, alopecia, or Graves' disease stable without systemic therapy for 2 years; hypothyroidism on hormone replacement; type 1 diabetes on insulin).

Transplantation History: Solid organ or hematopoietic stem cell transplantation.

Immunosuppressive Therapy:

Use of immunosuppressants (e.g., steroids) within 4 weeks before tumor sampling (Allowed: Physiologic glucocorticoid doses ≤12 mg/m²/day hydrocortisone equivalent; topical/nasal steroids).

Recent Anticancer Therapy:

Systemic anticancer treatment within 4 weeks before preconditioning (including investigational drugs; washout <5 half-lives if <4 weeks).

Planned participation in other interventional trials.

Active Infections:

HIV/syphilis antibody-positive; active HBV/HCV (Allowed: HBsAg/HBeAg+ if HBV DNA below LLN; HCV Ab+ if HCV RNA below LLN).

Active systemic infection or tuberculosis requiring treatment. Recent Surgery/Trauma: Major surgery or significant trauma within 4 weeks before screening; elective surgery planned during the study.

Poor Wound Healing: Surgery-related complications or delayed healing increasing risks of TIL therapy (per investigator judgment).

Other Malignancies: Additional primary malignancy within 5 years (Exceptions: Curatively treated basal/squamous cell carcinoma or carcinoma in situ).

Severe Respiratory Disease: History of severe ILD, COPD, pulmonary insufficiency, or symptomatic bronchospasm.

Gastrointestinal Complications: Surgical-required GI bleeding, bowel ischemia, or perforation.

CNS Involvement:

Leptomeningeal metastasis; uncontrolled/untreated CNS metastases (Exceptions: Asymptomatic lesions <1 cm, stable for ≥4 weeks without steroids/anticonvulsants).

Prior Cell Therapy: Previous treatment with similar cellular products. Pregnancy/Lactation: Pregnant or breastfeeding women.

Other Exclusions:

Psychiatric disorders, alcoholism, drug abuse, or other conditions deemed unsuitable by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AE) | 12 months
  To characterize the safety profile of HS-IT101 in patients with advanced solid tumor as assessed by incidence of adverse events
Serious Adverse Events (SAE) | 12 months
  To characterize the safety profile of HS-IT101 in patients with advanced solid tumor as assessed by incidence of serious adverse events
Objective Response Rate (ORR) | Up to 36 months
  To evaluate the efficacy of HS-IT101 in patients with advanced solid tumor, based on the objective response rate (ORR) as assessed by the Independent Review Committee (IRC) per RECIST v1.1
Time-to-response (TTR) | Up to 36 months
  To evaluate the efficacy of HS-IT101 in patients with advanced solid tumor by assessing the time-to-response (TTR) as assessed by the Investigator per RECIST v1.1
Duration of Response (DOR) | Up to 36 months
  To evaluate the efficacy of HS-IT101 in patients with advanced solid tumor by assessing the duration of response (DOR) as assessed by the Investigator per RECIST v1.1
Disease Control Rate (DCR) | Up to 36 months
  To evaluate the efficacy of HS-IT101 in patients with advanced solid tumor, based on the disease control rate (DCR) as assessed by the Independent Review Committee (IRC) per RECIST v1.1

SECONDARY OUTCOMES:
Progression-Free-Survival (PFS) | Up to 36 months
  To evaluate progression-free-survival (PFS) in patients with advanced solid tumor
Overall Survival (OS) | Up to 36 months
  To evaluate overall survival (OS) in patients with advanced solid tumor
Pharmacokinetic (PK) detection parameters for HS-IT101 | Up to 6 months
  peripheral blood lymphocyte subsets .
Pharmacokinetic (PK) detection parameters for HS-IT101 | Up to 6 months
  T-cell receptor (TCR) clonality

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No